CLINICAL TRIAL: NCT03555032
Title: A Phase I/II Study of the Safety and Efficacy of Talimogene Laherparepvec (T-VEC) Delivered by Intra-tumoural Injection in Combination With Isolated Limb Perfusion With Melphalan and Tumour Necrosis Factor-α in Patients With Advanced Extremity Tumours Including Metastatic Melanoma
Brief Title: TITAN (Tumoural Injection of T-VEC and Isolated Limb Perfusion)
Acronym: TITAN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4679
Record Dates: First submitted 2018-05-09; First posted 2018-06-13 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-03

CONDITIONS: Melanoma and Sarcoma
MeSH Terms: conditions — Melanoma; Sarcoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Intervention Model Description: Four Cohorts of patients staggered. Cohort 1: The first patient will need to be 30 days from the end of study treatment before patients can be consented to Cohort 2.
  Cohort 2: Assuming no Dose Limiting Toxicities in Cohort 1, two further patients will be recruited. Once these patients have passed 30 days from the end of study treatment Cohort 3 will open.
  Cohort 3: Three further patients will be recruited and be 30 days post before Cohort 4 opens.
  Cohort 4: Open recruitment for the remaining 9 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients will receive two pre-operative doses of T-VEC administered by intratumoural injection prior to a 3rd intratumoural dose given at the time of Isolated Limb Perfusion (ILP). No further treatment will be given.
  Interventions: Drug: Talimogene laherparepvec (T-VEC)

INTERVENTIONS:
Drug: Talimogene laherparepvec (T-VEC) — One dose of 1 x 106 PFU/mL. Two doses of 1 x 108 PFU/mL. Given by intra-tumoural (i.t.) injection.

SUMMARY:
This study will look at the safety and effects of combining a new drug called Talimogene Laherparepvec (T-VEC) with chemotherapy delivered by Isolated Limb Perfusion (ILP). The investigators want to find out whether these two treatments can be combined safely and whether T-VEC with ILP is better at treating your cancer than with ILP alone.

DETAILED DESCRIPTION:
This is a non-randomised, single-centre Phase I/II study of the combination of the oncolytic virus, TVEC, administered by intra-tumoural (i.t.) injection in combination with isolated limb perfusion with melphalan and tumour necrosis factor in patients with advanced extremity tumours.

The safety of T-VEC administered by i.t. injection followed by isolated limb perfusion will be assessed in an initial safety run in comprised of six subjects as described below.

Cohort 1: The first subject will be recruited and will receive an initial dose of T-VEC 4-6 weeks prior to isolated limb perfusion.

A further preoperative dose of i.t. T-VEC will be given at 2-3 weeks prior to isolated limb perfusion.

A third dose will be given on the day of isolated limb perfusion. Following isolated limb perfusion, no further doses of TVEC shall be given. No further patients will be recruited until this patient has passed 30 days from the end of the study treatment. If this patient experiences a dose limiting toxicity (DLT), the Trial Steering Committee (TSC) will meet to consider termination of the study.

Cohort 2: Assuming no DLTs in Cohort 1, two further patients will be recruited and receive the study treatment as described above. Once these patients have passed 30 days from the end of the study treatment, the TSC will meet and perform a safety assessment.

Cohort 3: Assuming TSC approval following Cohort 2, three further patients will be recruited and receive the study treatment as described above. Once these patients have passed 30 days from the end of the study treatment, the TSC will meet and perform a safety assessment.

Cohort 4: Open recruitment up to a maximum of 15 patients in total, unless otherwise indicated by the TSC.

If more than 1 DLT is observed at any point in the study, the Chief Investigator will notify the TSC and recruitment will be suspended until further notification from the TSC.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 years.
2. A confirmed histological diagnosis of in-transit malignant melanoma with or without regional lymph node metastases or limited visceral metastatic disease (AJCC Stage IIIb/c and IVa/b) or locally advanced soft-tissue sarcoma with or without regional or distant metastases (T2a/b, N0/1, M0/1) suitable for isolated limb perfusion.
3. Life expectancy of at least 3 months (as assessed, and documented by the Chief Investigator).
4. ECOG Performance Score of 0 to 2.
5. No continuing acute toxic effects of any prior radiotherapy, chemotherapy or surgical procedures, i.e., all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0) Grade 1.
6. Completed any previous chemotherapy at least 28 days before entry into the study.
7. Have baseline laboratory results as follows:

   * Absolute neutrophil count (ANC) 1.5 × 109 [SI units 109/L];
   * Platelets 100 ×109 [SI units 109/L] (without platelet transfusion);
   * Haemoglobin 9.0 g/dL [SI units gm/L] (with or without red blood cell (RBC) transfusion);
   * Serum creatinine 1.5 × upper limit of normal (ULN);
   * Bilirubin < 1.25 × ULN
   * ALT, AST and and alkaline phosphatase < 2 × ULN;
   * Calcium < 12 mg/dl (2.99 mmol/l).
8. Provide written informed consent in accordance with all applicable regulations and follow the study procedures. Patients must be capable

Exclusion Criteria:

1. Known cerebral metastases.
2. Have had concurrent immunotherapy during, and for the number of days equal to the half-life of that agent before or during, the study therapy.
3. Evidence of immunosuppression for any reason:

   * Known HIV disease
   * Acute or chronic hepatitis B or hepatitis C infection.
   * Chronic oral or systemic steroid medication use at a dose of > 10 mg/day of prednisolone or equivalent.
   * Other signs or symptoms of clinical immune system suppression.
4. Open herpetic skin lesions.
5. A history of hypersensitivity to T-VEC or its excipients.
6. Pregnant or breast-feeding female. Confirmation that women of childbearing potential are not pregnant with a negative serum and urine beta-human chorionic gonadotrophin (beta-hCG) pregnancy test results must be obtained within 7 days prior to treatment initiation (i.e. the 1st administration of T-VEC).
7. Fertile males and females who are unwilling to employ highly effective means of contraception during study treatment and for 3 months after the last dose of study treatment.
8. Previous treatment with T-VEC for active disease.
9. Require intermittent or chronic treatment with an anti-herpetic drug (e.g. acyclovir), other than intermittent topical use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The number of dose limiting toxicities and adverse events when T-VEC administered by intratumoural injection is combined with Isolated Limb Perfusion [Safety and Tolerability] | From first T-Vec administration to 52 week follow up.
  This will be assessed by serial blood tests and physical examinations from the first administration of T-VEC to 52 weeks follow-up
The percentage of patients achieving complete/partial response following treatment [Efficacy] | From T-Vec and ILP administration until 52 weeks follow up.
  This will be assessed by serial physical examinations and/or imaging from 4 weeks following therapy until 52 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hayes, Study Chair — The Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tulokas SKA, Kohtamaki LM, Makela SP, Juteau S, Alback A, Vikatmaa PJ, Mattila KE, Skytta TK, Koivunen JP, Tyynela-Korhonen K, Hernberg MM. Isolated limb perfusion with melphalan as treatment for regionally advanced melanoma of the limbs: results of 60 patients treated in Finland during 2007-2018. Melanoma Res. 2021 Oct 1;31(5):456-463. doi: 10.1097/CMR.0000000000000755. PMID 34132224